CLINICAL TRIAL: NCT05927064
Title: Multicenter Study Evaluating the Persistence, Efficacy and Tolerability of Methotrexate in Inflammatory Bowel Disease Patients
Brief Title: Study Evaluating the Persistence, Efficacy and Tolerability of Methotrexate in Inflammatory Bowel Disease Patients
Acronym: MICI-METHO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CARON Bénédicte, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2023PI032
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Methotrexate is one of the immunosuppressants used in chronic inflammatory bowel disease (IBD). It is indicated as monotherapy for induction and maintenance treatment of Crohn's disease (CD), or in combination with anti-tumor necrosis factor (TNF) agents for prevention of immunization.

The main objective is to assess the persistence rate of methotrexate treatment in patients followed for chronic inflammatory bowel disease (IBD).

DETAILED DESCRIPTION:
Methotrexate is one of the immunosuppressants used in chronic inflammatory bowel disease (IBD). It is indicated as monotherapy for induction and maintenance treatment of Crohn's disease (CD), or in combination with anti-tumor necrosis factor (TNF) agents for prevention of immunization Thiopurines are the most commonly used immunosuppressants in IBD, which contrasts with rheumatology data where methotrexate is the first-line immunosuppressant. Thiopurines and methotrexate have equivalent efficacy in CD 4.

Methotrexate is available in injectable (intramuscular (IM) or subcutaneous (SC)) or tablet form. In IBD, only parenteral administration has been shown to be effective. There is no consensus on the optimal maintenance dosage.

Tolerance problems remain an obstacle to its use, even if the side effects are not severe.

In this context, the objectives of this study are to describe the use of methotrexate in current practice in patients followed for IBD, its persistence, compliance, tolerance, as well as the factors associated with the persistence of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Person who has received full information on the organization of the research and has not objected to the use of this data
2. Age ≥18 years
3. Certain diagnosis of IBD (European Crohn's Colitis Organization criteria)
4. Introduction of methotrexate mono- or combination therapy between January 1, 2015 and December 31, 2022
5. Minimum 6-month follow-up after initiation of methotrexate therapy
6. Person affiliated with a social security plan or beneficiary of such a plan

Exclusion Criteria:

1. Age <18 years
2. Person referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code

   * Pregnant woman, parturient or nursing mother
   * Minor (not emancipated)
   * Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
   * A person of full age who is unable to give consent
3. Persons deprived of liberty by a judicial or administrative decision, persons under psychiatric care by virtue of articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients followed for IBD treated with methotrexate between 01/01/2015 and 12/31/2022.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Persistence rate of methotrexate treatment in chronic inflammatory bowel disease patients | minimum follow-up of 6 months post-induction of treatment and maximum on the date of cessation of treatment or date of last news 12/31/2022
  Persistence is measured as the time between starting treatment and stopping the drug or switching to another drug.

SECONDARY OUTCOMES:
Assess the effectiveness of induction therapy with methotrexate for Crohn's patient | minimum follow-up of 6 months post-induction of treatment and maximum on the date of cessation of treatment or date of last news 12/31/2022
  Clinical response defined as a decrease of at least 3 points in the Harvey-Bradshaw Index (HBI) for CD assessed at 6 months of methotrexate therapy.
  The Harvey-Bradshaw Index consists of a few questions (n=5) to quickly categorize the severity of Crohn's disease and detect remission.
  Harvey-Bradshaw Index Score:
  Remission: <5 Mild Disease: 5 to 7 Moderate Disease: 8 to 16 Severe Disease: >16
Assess the effectiveness of induction therapy with methotrexate for Ulcerative colitis patient | minimum follow-up of 6 months post-induction of treatment and maximum on the date of cessation of treatment or date of last news 12/31/2022
  Clinical response defined as a decrease of at least 3 points in the partial Mayo score for Ulcerative colitis (UC) assessed at 6 months of methotrexate therapy
  Mayo score composed by 4 items: stool frequency; rectal bleeding, mucosal appearance at endoscopy and physician rating of disease activity.
  Mayo score:
  Score <2 : no activity Score between 3 and 5: mild activity Score between 6 and 10 :moderate activity Score >11 : severe activity
Assess the safety of methotrexate therapy | minimum follow-up of 6 months post-induction of treatment and maximum on the date of cessation of treatment or date of last news 12/31/2022
  Adverse reactions associated with methotrexate treatment: hematological, hepatic, pulmonary, renal toxicity, allergic reaction, abdominal pain, nausea, vomiting.
Describe the reasons for discontinuation of methotrexate therapy | minimum follow-up of 6 months post-induction of treatment and maximum on the date of cessation of treatment or date of last news 12/31/2022
  Reasons for discontinuing methotrexate: inefficiency and intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte CARON, MD, Principal Investigator — CHRU of Nancy, Hepatogastroenterology Department
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Feagan BG, Rochon J, Fedorak RN, Irvine EJ, Wild G, Sutherland L, Steinhart AH, Greenberg GR, Gillies R, Hopkins M, et al. Methotrexate for the treatment of Crohn's disease. The North American Crohn's Study Group Investigators. N Engl J Med. 1995 Feb 2;332(5):292-7. doi: 10.1056/NEJM199502023320503. PMID 7816064
- [Result] Mate-Jimenez J, Hermida C, Cantero-Perona J, Moreno-Otero R. 6-mercaptopurine or methotrexate added to prednisone induces and maintains remission in steroid-dependent inflammatory bowel disease. Eur J Gastroenterol Hepatol. 2000 Nov;12(11):1227-33. doi: 10.1097/00042737-200012110-00010. PMID 11111780
- [Result] Nielsen OH, Ainsworth MA, Steenholdt C. Methotrexate for inflammatory bowel disease: time for reconsideration. Expert Rev Gastroenterol Hepatol. 2019 May;13(5):407-409. doi: 10.1080/17474124.2019.1596797. Epub 2019 Mar 21. No abstract available. PMID 30895827
- [Result] Ardizzone S, Bollani S, Manzionna G, Imbesi V, Colombo E, Bianchi Porro G. Comparison between methotrexate and azathioprine in the treatment of chronic active Crohn's disease: a randomised, investigator-blind study. Dig Liver Dis. 2003 Sep;35(9):619-27. doi: 10.1016/s1590-8658(03)00372-4. PMID 14563183